CLINICAL TRIAL: NCT07336342
Title: Mindfulness-based Cognitive Therapy for the Chronic Pain-depression Co-morbidity Among Older Black Adults in the Community; The Quiet Focus Open Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Tony V. Pham, MD, Principal Investigator and Psychiatrist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024P001995; K23AT012363 (NIH)
Record Dates: First submitted 2026-01-08; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-09

CONDITIONS: Chronic Pain; Depression
Keywords: mindfulness-based cognitive therapy; mind-body; chronic pain; depression; older adult
MeSH Terms: conditions — Chronic Pain; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Quiet Focus (Experimental)
  Interventions: Behavioral: Quiet Focus

INTERVENTIONS:
Behavioral: Quiet Focus — Mindfulness-based cognitive therapy adapted for older adults at-risk for chronic pain and depression.

SUMMARY:
The goal of this clinical trial is to pilot an adaptation of mindfulness-based cognitive therapy for chronic pain and depression. The main questions it aims to answer in a later fully powered randomized controlled trial are:

* Is an adaptation of mindfulness-based cognitive therapy for older Black adults able to improve quality of life?
* Will an adapted mindfulness based cognitive therapy reduce pain interference to a greater degree than a traditional health enhancement program?

DETAILED DESCRIPTION:
Co-morbid chronic pain-depression is common among older Black adults and this co-morbidity worsens physical and emotional function. Access to evidence based non-pharmacological management is limited. Mindfulness based cognitive therapy (MBCT) is an evidence-based, non-pharmacological intervention that could address the chronic pain-depression co-morbidity among older Black adults, but it requires tailoring. The proposed study will establish the feasibility, acceptability and credibility of Quiet Focus, a cultural adaptation of MBCT aimed at the chronic pain-depression co-morbidity among older Black adults in the community.

ELIGIBILITY:
Participant Inclusion Criteria

1. Older adult (age ≥ 50)
2. All individuals who identify with one or more nationalities or ethnic groups originating in any of the Black racial groups of Africa
3. Pain in muscles, joints, bones, or associated soft tissues (NRS>4) lasting longer than 3 months
4. Depressed (PHQ-9 score of 5-14)
5. English fluency/literacy
6. Ability and willingness to participate via in-person and video
7. No change to type or dose of antidepressant medications for at least 6 weeks prior to screening
8. Willing to provide informed consent and comply with all aspects of the protocol

Participant Exclusion Criteria

1. Moderately severe or severe depressive symptoms (PHQ-9 ≥ 15)
2. Current substance abuse/dependence
3. Significant cognitive impairment
4. History of more than 8 sessions of cognitive-behavioral therapy
5. History of previous training in mindfulness or undergoing counseling more than once a month
6. History of or current diagnosis of psychosis
7. Active suicidal ideation (PHQ-9 item #9 or otherwise reported during screening) or self-harm within the past 90 days
8. Current participation in another behavioral clinical trial

Ages: 50 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
The Credibility and Expectancy Questionnaire | From enrollment to 3 months from the end of treatment at 8 weeks
  This scale measures participant expectations around the study's positive outcomes, with measures ranging from 0 (not at all expected) to 9 (extremely expected). A higher score indicate greater trust in the study design and an openness to potential benefits.
The Client Satisfaction Questionnaire | Administered at the end of treatment at 8 weeks and at the three month follow up visit.
  Three item scale measuring patient satisfaction with the program. Scores for each item range from 1 (unsatisfied) to 4 (very satisfied).
Modified Patient Global Impression of Change | At end of 8 week program (post test) and again at 3 month follow up visit.
  Measures participant impressions of overall change with one being very much improved and eight being very much worse. Lower scores indicate improvement.

SECONDARY OUTCOMES:
Numerical Rating Scale | From enrollment to 3 months from the end of treatment at 8 weeks.
  Numerical rating of pain with lower scores indicating less pain overall (0 = no pain) and higher scores indicating more pain (10 = worst ever pain) over the past week.
PROMIS Physical Function | From enrollment to 3 months from the end of treatment at 8 weeks
  The PROMIS Depression raw score is calculated by summing item responses, each rated on a 5-point Likert scale where 1 = "Never" and 5 = "Always," with higher scores indicating more severe depressive symptoms. This raw score is converted to a T-score using a standardized table, where 50 represents the average level in the general population and 10 is the standard deviation.
PROMIS Anxiety | From enrollment to 3 months from the end of treatment at 8 weeks
  The PROMIS Anxiety raw score is calculated by summing item responses, each rated on a 5-point Likert scale where 1 = "Never" and 5 = "Always," with higher scores reflecting greater anxiety symptoms. The raw score is then converted to a T-score using a standardized scoring table, with 50 representing the population average and 10 as the standard deviation.
PROMIS Depression | From enrollment to 3 months from the end of treatment at 8 weeks
  The PROMIS Depression raw score is calculated by summing item responses, each rated on a 5-point Likert scale where 1 = "Never" and 5 = "Always," with higher scores indicating more severe depressive symptoms. This raw score is converted to a T-score using a standardized table, where 50 represents the average level in the general population and 10 is the standard deviation.
PROMIS Emotional Support | From enrollment to 3 months from the end of treatment at 8 weeks.
  The PROMIS Emotional Support raw score is calculated by summing item responses, each rated on a 5-point Likert scale where 1 = "Never" and 5 = "Always," with higher scores indicating greater perceived emotional support. This raw score is converted to a T-score using a standardized table, where 50 represents the average for the general population and 10 is the standard deviation.
Measure of Current Status Part A | From enrollment to 3 months from the end of treatment at 8 weeks
  The Measure of Current Status Part A (MOCS-A) is a self-report questionnaire that measures ability to manage stress. The score is calculated by summing responses to each item, rated on a 5-point Likert scale where 0 = "I cannot do this at all" and 4 = "I can do this extremely well," with higher scores reflecting greater confidence in coping skills. The scale measures current perceived ability to manage stress across areas like relaxation, awareness of tension, assertiveness, and coping confidence.
Cognitive and Affective Mindfulness Scale-Revised | From enrollment to 3 months from the end of treatment at 8 weeks
  Description: The Cognitive and Affective Mindfulness Scale - Revised (CAMS-R) measures percieved ability to complete mindfulness tasks such as meditation, with a 0 being rarely/not at all and a 3 being almost always. Higher scores indicate greater ability to practice mindfulness skills.
Chronic Pain Acceptance Questionnaire | From enrollment to 3 months from the end of treatment at 8 weeks
  The Chronic Pain Acceptance Questionnaire (CPAQ)*= raw score is calculated by summing responses to each item, rated on a 7-point Likert scale where 0 = "Never true" and 6 = "Always true," with higher scores indicating greater acceptance of chronic pain. The scale assesses two key areas: pain willingness(the ability to experience pain without trying to control or avoid it) and activity engagement (continuing meaningful activities despite pain).
Pain Self-Efficacy Questionnaire | From enrollment to 3 months from the end of treatment at 8 weeks
  The Pain Self-Efficacy Questionnaire (PSEQ) measures confidence in engaging in activities despite chronic pain. Higher scores indicate greater confidence (6 = complete confidence) and lower scores indicate lower confidence (0 = not at all confident).
Pain Catastrophizing Scale | From enrollment to 3 months from the end of treatment at 8 weeks
  The Pain Catastrophizing Scale (PCS) score is calculated by summing responses to each item, rated on a 5-point Likert scale where 0 = "Not at all" and 4 = "All the time," with higher scores indicating greater levels of catastrophic thinking related to pain. The scale measures three components of pain catastrophizing: rumination, magnification, and helplessness.
Tampa Kinesiophobia Scale | From enrollment to 3 months from the end of treatment at 8 weeks
  The Tampa Kinesiophobia Scale (TKS) measures fear of movement and is calculated by summing responses to each item, rated on a 4-point Likert scale where 1 = "Strongly disagree" and 4 = "Strongly agree," with higher scores indicating greater fear of movement or reinjury due to physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Tony V Pham, MD, MScGH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the trial.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

DOCUMENTS (1):
  • Informed Consent Form (2024-07-25): https://cdn.clinicaltrials.gov/large-docs/42/NCT07336342/ICF_000.pdf